CLINICAL TRIAL: NCT00456599
Title: A Multi-Institutional Phase II Study of Neoadjuvant Gemcitabine and Oxaliplatin With Radiation Therapy in Patients With Pancreatic Cancer
Brief Title: Study of Gemcitabine and Oxaliplatin With Radiation Therapy in Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Sanofi (Industry); Johns Hopkins University (Other); Princess Margaret Hospital, Canada (Other); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2006.025; HUM 4531 (Other: University of Michigan IRBMED); NCT00426738 (obsolete NCT alias)
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin & gemcitabine with radiation (Experimental): This study will examine a sequence of treatments including pre-operative chemotherapy and radiation, surgery and post-operative chemotherapy for resectable pancreatic cancer.
  Interventions: Drug: gemcitabine; Drug: oxaliplatin; Procedure: Radiation

INTERVENTIONS:
Drug: gemcitabine — Gemcitabine 1000mg/m2 will be infused over 30 minutes on days 1, 8, and 15 of a treatment cycle.
  Other Names: Gemzar
Drug: oxaliplatin — Oxaliplatin 85mg/m2 will be infused following gemcitabine over approximately 90 minutes on days 1 and 15 of a treatment cycle.
  Other Names: Eloxatin
Procedure: Radiation — The total dose in a three week treatment block will be 30 Gy in 2.0 Gy fractions.
  Other Names: RT

SUMMARY:
This study will examine a sequence of treatments including pre-operative chemotherapy and radiation, surgery and post-operative chemotherapy for resectable pancreatic cancer.

DETAILED DESCRIPTION:
This study will examine a sequence of treatments including pre-operative chemotherapy and radiation, surgery and post-operative chemotherapy for resectable pancreatic cancer. This research treatment will evaluate the combination of two chemotherapy agents, oxaliplatin and gemcitabine with radiation therapy. The researchers have already done studies using oxaliplatin, gemcitabine and radiation therapy together for pancreatic cancer. They want to build on the information they have from this previous research and do the research at multiple sites. They will use this study to determine how well people do who are treated with gemcitabine, oxaliplatin, and radiation therapy prior to having surgery for their pancreatic cancer. The researchers will also gather more information about what type of side effects occur with this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytologic or histologic confirmation of carcinoma arising in the pancreas.
* Patients must be deemed resectable or borderline resectable based on criteria in section 4.2 prior to registration.
* Patients must have an expected life expectancy of at least 12 weeks and a Zubrod performance status of < 2.
* Patients must have adequate organ function defined as follows: absolute neutrophil count of > 1500/mm3, platelets > 100,000/mm3, serum Cr < 1.5 mg/dl, total bilirubin < 3.0 mg/dl with relief of biliary obstruction if present (PTC tube or endobiliary stent).
* Patients must be free of other active systemic malignancy, ongoing infection, including HIV infection, or any other serious uncontrolled, concomitant systemic disorders or psychiatric condition that would interfere with the safe delivery of protocol therapy.
* Patients must be aware of the investigational nature of the therapy and provide written informed consent.
* Patients must have no history of previous chemotherapy for pancreatic cancer or any abdominal radiation therapy.
* Patients must not have used any investigational agent in the month before enrollment into the study.

Exclusion Criteria:

* Patients with neuroendocrine tumors are excluded.
* Patients with preexisting peripheral neuropathy > grade 2 are ineligible.
* Pregnant or nursing women are ineligible and patients of reproductive potential must agree to use an effective contraceptive method during participation in this trial and for 6 months after trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-04; Primary Completion 2012-05 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, MD, Principal Investigator — University of Michigan
Locations (4):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Ohio State University, Columbus, Ohio
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Kim EJ, Ben-Josef E, Herman JM, Bekaii-Saab T, Dawson LA, Griffith KA, Francis IR, Greenson JK, Simeone DM, Lawrence TS, Laheru D, Wolfgang CL, Williams T, Bloomston M, Moore MJ, Wei A, Zalupski MM. A multi-institutional phase 2 study of neoadjuvant gemcitabine and oxaliplatin with radiation therapy in patients with pancreatic cancer. Cancer. 2013 Aug 1;119(15):2692-700. doi: 10.1002/cncr.28117. Epub 2013 May 29. PMID 23720019

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine and Oxaliplatin With Radiation Therapy: Gemcitabine and Oxaliplatin with radiation therapy in localized pancreatic cancer.
Period: Overall Study
Arm/Group | Gemcitabine and Oxaliplatin With Radiation Therapy
Started | 71
Completed Cycle 1 | 66 (Of the 71 patients, 1 was removed for noncompliance; 2 withdrew; 2 did not complete cycle 1.)
Initiated Cycle 2 | 61 (5 patients were removed from study prior to initiation of a second cycle.)
Completed Protocol Surgery | 48 (Forty-eight patients (71%) underwent laparotomy according to the protocol.)
Completed Resection | 43 (43 patients underwent resection.)
Post-Surgery Adjuvent Therapy | 26 (After resection, 26 patients (68%) initiated adjuvant therapy.)
Completed 4th Cycle of Chemotherapy | 24 (24 patients (63%) completed a fourth cycle of chemotherapy.)
Completed | 68
Not Completed | 3
Not completed — Non-compliance | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 68 patients were evaluable. 71 patients were enrolled however 1 was removed from study during cycle 1 due to non-compliance and 2 additional patients withdrew for reasons not related to toxicity or progression.
Groups:
- Oxaliplatin & Gemcitabine With Radiation: Protocol treatment consisted of four 28 day cycles of chemotherapy: 2 cycles before surgery and 2 cycles before surgery and 2 cycles after. Gemcitabine (1 g/m2 infused over 30 minutes) was administered on days 1, 8, and 15 of each cycle; oxaliplatin (85 mg/m2 infused over 90 minutes) was administered on days 1 and 15. Radiation therapy was delivered concurrently with the first cycle of chemotherapy in 2-Gray [Gy] fractions (total dose, 30 Gy).
Arm/Group | Oxaliplatin & Gemcitabine With Radiation
Number analyzed (Participants) | 68
Age, Continuous [Mean (Full Range); unit: years] | 64 [42 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 58
  Canada | 10

OUTCOME MEASURES:

1. Primary Outcome: Two-year Disease Free Survival.
Description: The percent of patients alive and disease-free at two years.
Time Frame: two years
Population: 43 patients underwent resection. 41 of the 43 had R0/R1 (surgical margin status) resection. Patients with R02 surgical margins (portions of the tumor visible to the naked eye were not removed) were not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Oxaliplatin & Gemcitabine With Radiation
Number analyzed (Participants) | 41
percentage of patients | 26.1 [16.1 to 37.4]

2. Secondary Outcome: Time to Treatment Failure
Description: Median time for disease recurrence after surgery.
Time Frame: 2 years
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Oxaliplatin & Gemcitabine With Radiation
Number analyzed (Participants) | 41
months | 10.4 [2.3 to 35.8]

3. Secondary Outcome: Overall Survival
Description: Percent overall survival was calculated for all evaluable patients.
Time Frame: 5 years
Population: Of the 71 eligible patients, 68 were evaluable for overall response (1 patient was removed from study during cycle 1 for noncompliance, and 2 additional patients withdrew for reasons not related to toxicity or progression).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oxaliplatin & Gemcitabine With Radiation
Number analyzed (Participants) | 68
months | 18.2 [13 to 26.9]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were captured on day 1 until 30 days post treatment.
Arm/Group | Oxaliplatin & Gemcitabine With Radiation
Serious Adverse Events (participants affected / at risk) | 28/71
Other Adverse Events (participants affected / at risk) | 57/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin & Gemcitabine With Radiation (N=71)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (2)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 2 (2)
Creatine phosphokinase increased (Investigations) | 1 (1)
Death (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
GI - Other (Specify) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
General symptom (General disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Hepatobiliary - Other (Specify) (Hepatobiliary disorders) | 1 (2)
Hyperbilirubinemia (Investigations) | 1 (1)
Infection, Biliary tree (Infections and infestations) | 1 (3)
Leukocytes (Investigations) | 5 (8)
Leukopenia (Investigations) | 4 (8)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lymph leakage (Vascular disorders) | 1 (1)
Lymphopenia (Investigations) | 5 (7)
Nausea (Gastrointestinal disorders) | 3 (4)
Neutrophil count decreased (Investigations) | 6 (10)
Neutrophils (Investigations) | 2 (4)
Opportunisitic infection (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 3 (5)
Platelets (Investigations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin & Gemcitabine With Radiation (N=71)
Constipation (Gastrointestinal disorders) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 8 (10)
Fatigue (General disorders) | 15 (29)
Hemoglobin (Blood and lymphatic system disorders) | 15 (59)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (6)
Hyperbilirubinemia (Investigations) | 6 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 (23)
Hypokalemia (Metabolism and nutrition disorders) | 5 (6)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Leukocytes (Blood and lymphatic system disorders) | 26 (59)
Leukopenia (Investigations) | 9 (10)
Lymphopenia (Investigations) | 16 (26)
Nausea (Gastrointestinal disorders) | 15 (20)
Neutrophil count decreased (Investigations) | 9 (13)
Neutrophils (Investigations) | 22 (53)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5)
Platelet count decreased (Investigations) | 13 (17)
Platelets (Investigations) | 29 (70)
Taste alteration (Nervous system disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 8 (10)
Weight loss (Metabolism and nutrition disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No